CLINICAL TRIAL: NCT03891758
Title: Phase 3 Study of BK1310 Compared With ActHIB® and Tetrabik in Healthy Infants: A Randomized, Assessor-blind, Active-controlled
Brief Title: Confirmatory Study of BK1310 in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: The Research Foundation for Microbial Diseases of Osaka University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BK1310-J03; jRCT2080224611 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2019-03-24; First posted 2019-03-27 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Tetanus; Diphtheria; Pertussis; Poliomyelitis; Bacterial Meningitis
Keywords: Haemophilus influenza type b; Adsorbed Diphtheria-purified Pertussis-Tetanus- Inactivate poliovirus combined vaccine; Hib; DPT-IPV
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough; Poliomyelitis; Meningitis, Bacterial; Haemophilus Infections | interventions — HibTITER protein, Haemophilus influenzae; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BK1310 (Experimental)
  Interventions: Biological: DPT-IPV-Hib
- ActHIB® and Tetrabik (Active Comparator)
  Interventions: Biological: Hib vaccine; Biological: DPT-IPV

INTERVENTIONS:
Biological: DPT-IPV-Hib — 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
  Other Names: BK1310
  Arms: BK1310
Biological: Hib vaccine — 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
  Other Names: ActHIB®
  Arms: ActHIB® and Tetrabik
Biological: DPT-IPV — 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
  Other Names: Tetrabik
  Arms: ActHIB® and Tetrabik

SUMMARY:
The purpose of this study is to evaluate immunogenicity of BK1310 for all antigens (anti-PRP, diphtheria toxin, pertussis, tetanus toxin, and polio virus), after 3 times of injection, when compared noninferiority with co-administration of ActHIB® and Tetrabik, as well as efficacy and safety, in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged ≥2 and <43 months at the first vaccination of the study drug (recommended: ≥2 and <7 months)
* Written informed consent is obtained from a legal guardian (parent)

Exclusion Criteria:

* Possibility of anaphylaxis due to food or pharmaceuticals
* With experience of Hib infection, diphtheria, pertussis, tetanus or acute poliomyelitis
* With experience of Hib, diphteria, pertussis, tetanus or polio vaccination.
* Participated in other studies within 12 weeks before obtaining consent
* Considered to be not eligible by the principal investigators (sub-investigators) of the enrollment

Additional screening criteria check may apply for qualification.

Ages: 2 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational Site, Fukuoka, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nakano T, Hasegawa M, Endo M, Matsuda K, Tamai H. Immunogenicity and safety of adsorbed diphtheria-purified pertussis-tetanus-inactivated polio (Sabin strain)-Haemophilus type b conjugate combined vaccine (DPT-IPV-Hib) in healthy Japanese Infants >/= 2 and < 43 months of Age: A phase III, multicenter, active controlled, assessor-blinded, randomized, parallel-group study. Vaccine. 2024 Apr 30;42(12):3134-3143. doi: 10.1016/j.vaccine.2023.03.077. Epub 2024 Apr 6. PMID 38582691

RESULTS

PARTICIPANT FLOW:
Groups:
- BK1310: DPT-IPV-Hib (Combined Vaccine) 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
- ActHIB® and Tetrabik (Control): Hib vaccine and DPT-IPV 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
Period: Overall Study
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Started | 133 | 134
Completed | 131 | 132
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by parent/guardian | 0 | 2

BASELINE CHARACTERISTICS:
Population: Excluding 1 subject(control: 1 subject) whose all antibody titers could not be measured at Visit 4
Groups:
- Total: Total of all reporting groups
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control) | Total
Number analyzed (Participants) | 133 | 133 | 266
Age, Customized [Count of Participants; unit: Participants]
  >=2 and <3 months | 124 | 125 | 249
  >=3 months | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 62 | 135
  Male | 60 | 71 | 131
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 133 | 133 | 266

OUTCOME MEASURES:

1. Primary Outcome: Antibody Prevalence Rate Against Anti-PRP With 1 μg/mL or Higher, Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus, Defined as the Percentage of Participants With the Antibody Against Anti-PRP
Description: Antibody prevalence rate is defined as the percentage of participants whose criteria of each antibody titer: Anti-diphtheria antibody concentrations: >=0.1 IU/mL, Anti-PT antibody concentrations: >=10.0 EU/mL, Anti-FHA antibody concentrations: >=10.0 EU/mL, Anti-tetanus antibody concentrations: >=0.01 IU/mL, Anti-poliovirus serotype 1,2 and 3 antibody titers (fold) >=8
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 267 to 266. Control group: due to withdrawal by parent/guardian (n=1) . In BK1310 group number of subjects further decreased due to insufficient sample volume (polio serotype1,2 and 3: n=2 each). In control group number of subjects further decreased due to insufficient sample volume (polio serotype1,2 and 3: n=1 each).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 133 | 133
percentage of participants
  Antibody prevalence rate against anti-PRP with 1 μg/mL or higher | 100.0 [97.3 to 100.0] | 88.7 [82.1 to 93.5]
  Antibody prevalence rate against diphtheria toxin | 99.2 [95.9 to 100.0] | 98.5 [94.7 to 99.8]
  Antibody prevalence rate against pertussis （PT） | 100.0 [97.3 to 100.0] | 100.0 [97.3 to 100.0]
  Antibody prevalence rate against pertussis (FHA) | 100.0 [97.3 to 100.0] | 100.0 [97.3 to 100.0]
  Antibody prevalence rate against tetanus toxin | 100.0 [97.3 to 100.0] | 99.2 [95.9 to 100.0]
  Antibody prevalence rate against polio virus serotype 1: number analyzed (Participants) | 131 | 132
  Antibody prevalence rate against polio virus serotype 1 | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Antibody prevalence rate against polio virus serotype 2: number analyzed (Participants) | 131 | 132
  Antibody prevalence rate against polio virus serotype 2 | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Antibody prevalence rate against polio virus serotype 3: number analyzed (Participants) | 131 | 132
  Antibody prevalence rate against polio virus serotype 3 | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]

2. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 267 to 266. Control group: due to withdrawal by parent/guardian (n=1) .
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 133 | 133
percentage of participants | 100.0 [97.3 to 100.0] | 100.0 [97.3 to 100.0]

3. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4weeks after the primary immunization (Visit 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 133 | 133
µg/mL | 23.688 [20.208 to 27.768] | 6.698 [5.357 to 8.374]

4. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 1 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 4, number of subjects decreased from 267 to 266. Control group: due to withdrawal by parent/guardian (n=1) .
  For antibody analysis at Visit 6, number of subjects decreased from 266 to 264. BK1310 group: due to Adverse event (n=2, onty 1 patient was able to collect a sample at discontinuation. The data at this time point was included in Visit 6). Control group: due to withdrawal by parent/guardian (n=1) .
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 132 | 132
percentage of participants | 100.0 [97.2 to 100.0] | 98.5 [94.6 to 99.8]

5. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 132 | 132
percentage of participants | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]

6. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 132 | 132
µg/mL | 56.545 [47.963 to 66.661] | 34.246 [28.835 to 40.672]

7. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 133 | 133
IU/mL | 1.841 [1.533 to 2.211] | 1.283 [1.050 to 1.567]

8. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 133 | 133
EU/mL
  pertussis （PT） | 155.30 [141.53 to 170.41] | 200.24 [183.42 to 218.61]
  pertussis （FHA） | 56.48 [51.07 to 62.46] | 85.24 [76.96 to 94.40]

9. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 133 | 133
IU/mL | 0.473 [0.408 to 0.548] | 0.158 [0.124 to 0.203]

10. Secondary Outcome: Geometric Mean Antibody Titer Against Polio Virus
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 131 | 132
IU/mL
  polio virus serotype 1 | 684.95 [539.57 to 869.49] | 663.98 [512.66 to 859.96]
  polio virus serotype 2 | 2026.44 [1733.39 to 2369.04] | 1767.97 [1498.47 to 2085.94]
  polio virus serotype 3 | 1729.00 [1487.12 to 2010.23] | 2075.06 [1777.90 to 2421.90]

11. Secondary Outcome: Antibody Prevalence Rate Against Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus, Defined as the Percentage of Participants With the Antibody Against Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus
Description: as for outcome 1
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 4, number of subjects decreased from 267 to 266. Control group: due to withdrawal by parent/guardian (n=1). For antibody analysis at Visit 6, number of subjects decreased from 266 to 264. BK1310 group: due to Adverse event (n=2). Control group: due to withdrawal by parent/guardian (n=1) .In BK1310 group number of subjects further decreased due to insufficient sample volume (tetanus: n=1, polio serotype1,2 and 3: n=1 each).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 132 | 132
percentage of participants
  Antibody prevalence rate against diphtheria toxin | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Antibody prevalence rate against pertussis （PT） | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Antibody prevalence rate against pertussis （FHA） | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Antibody prevalence rate against tetanus toxin: number analyzed (Participants) | 131 | 132
  Antibody prevalence rate against tetanus toxin | 100.0 [97.2 to 100.0] | 99.2 [95.9 to 100.0]
  Antibody prevalence rate against polio virus serotype 1: number analyzed (Participants) | 131 | 132
  Antibody prevalence rate against polio virus serotype 1 | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Antibody prevalence rate against polio virus serotype 2: number analyzed (Participants) | 131 | 132
  Antibody prevalence rate against polio virus serotype 2 | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Antibody prevalence rate against polio virus serotype 3: number analyzed (Participants) | 131 | 132
  Antibody prevalence rate against polio virus serotype 3 | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]

12. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 132 | 132
IU/mL | 9.766 [8.758 to 10.890] | 8.961 [8.035 to 9.994]

13. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 132 | 132
EU/mL
  Geometric mean antibody titer against pertussis （PT） | 209.05 [189.40 to 230.74] | 279.62 [254.28 to 307.49]
  Geometric mean antibody titer against pertussis （FHA） | 144.73 [128.04 to 163.59] | 221.34 [194.79 to 251.51]

14. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 4, number of subjects decreased from 267 to 266. Control group: due to withdrawal by parent/guardian (n=1) . For antibody analysis at Visit 6, number of subjects decreased from 266 to 264. BK1310 group: due to Adverse event (n=2). Control group: due to withdrawal by parent/guardian (n=1) .In BK1310 group number of subjects further decreased due to insufficient sample volume (n=1).
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 131 | 132
IU/mL | 1.904 [1.595 to 2.272] | 0.598 [0.457 to 0.783]

15. Secondary Outcome: Fold Change in Geometric Mean Antibody Titer Against Polio Virus
Time Frame: Baseline and 4 weeks after the primary immunization (Visit 6)
Population: For antibody analysis at Visit 4, number of subjects decreased from 267 to 266. Control group: due to withdrawal by parent/guardian (n=1) . For antibody analysis at Visit 6, number of subjects decreased from 266 to 264. BK1310 group: due to Adverse event (n=2). Control group: due to withdrawal by parent/guardian (n=1) .In BK1310 group number of subjects further decreased due to insufficient sample volume (polio serotype1,2 and 3: n=1 each).
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 131 | 132
fold change
  Geometric mean antibody titer against polio virus serotype 1 | 2524.05 [2110.26 to 3018.98] | 2662.91 [2254.04 to 3145.95]
  Geometric mean antibody titer against polio virus serotype 2 | 8821.88 [7678.48 to 10135.54] | 7512.10 [6425.09 to 8783.01]
  Geometric mean antibody titer against polio virus serotype 3 | 6439.23 [5472.88 to 7576.21] | 7355.96 [6324.16 to 8556.09]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | BK1310 | ActHIB® and Tetrabik (Control)
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/134
Serious Adverse Events (participants affected / at risk) | 9/133 | 11/134
Other Adverse Events (participants affected / at risk) | 131/133 | 132/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BK1310 (N=133) | ActHIB® and Tetrabik (Control) (N=134)
Cholangiectasis congenital (Congenital, familial and genetic disorders) | 0 | 1
Adenovirus infection (Infections and infestations) | 1 | 1
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fractured skull depressed (Injury, poisoning and procedural complications) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Kawasaki's disease (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BK1310 (N=133) | ActHIB® and Tetrabik (Control) (N=134)
Crying (General disorders) | 37 | 38
Injection site erythema (General disorders) | 105 | 107
Injection site induration (General disorders) | 63 | 72
Injection site pain (General disorders) | 18 | 26
Injection site swelling (General disorders) | 41 | 47
Irritability postvaccinal (General disorders) | 40 | 46
Pyrexia (General disorders) | 91 | 88
Bronchitis (Infections and infestations) | 19 | 18
Conjunctivitis (Infections and infestations) | 7 | 6
Gastroenteritis (Infections and infestations) | 8 | 8
Nasopharyngitis (Infections and infestations) | 39 | 38
Otitis media (Infections and infestations) | 8 | 7
Pharyngitis (Infections and infestations) | 7 | 7
Upper respiratory tract infection (Infections and infestations) | 23 | 21
Decreased appetite (Metabolism and nutrition disorders) | 21 | 23
Hypersomnia (Nervous system disorders) | 36 | 31
Insomnia (Psychiatric disorders) | 24 | 28
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 13 | 17
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 | 11
Eczema (Skin and subcutaneous tissue disorders) | 13 | 17
Eczema infantile (Skin and subcutaneous tissue disorders) | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03891758/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT03891758/SAP_001.pdf